CLINICAL TRIAL: NCT06435026
Title: Optimizing PrEP Regimens for Pregnant Women in Sub-Saharan Africa (O-PrEP Study) - Stage 1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-2056; R01AI157859 (NIH)
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: HIV; Prevention; Pregnancy
Keywords: HIV; PrEP; Pregnancy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard Dose (Other): daily oral FTC/TDF standard dose (200mg/300mg, n=18)
  Interventions: Drug: FTC/TDF 200mg/300mg
- 150% standard dose (Other): daily oral FTC/TDF dose (300mg/450mg, n=18),
  Interventions: Drug: FTC/TDF 300mg/450mg
- 200% standard dose (Other): daily oral FTC/TDF (400mg/600mg, n=18)
  Interventions: Drug: FTC/TDF 400mg/600mg

INTERVENTIONS:
Drug: FTC/TDF 200mg/300mg — Standard Dose
  Other Names: PrEP
  Arms: Standard Dose
Drug: FTC/TDF 300mg/450mg — 150% Standard Dose
  Other Names: PrEP
  Arms: 150% standard dose
Drug: FTC/TDF 400mg/600mg — 200% Standard Dose
  Other Names: PrEP
  Arms: 200% standard dose

SUMMARY:
This study aims: (1) to determine the optimal dose of emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) for daily oral pre-exposure prophylaxis (PrEP) during pregnancy based on drug pharmacokinetics, and (2) evaluate the maternal and infant safety of increased FTC/TDF doses during these periods.

DETAILED DESCRIPTION:
This is a staged study to assess the pharmacokinetics (PK) and safety of increased FTC/TDF doses for PrEP during pregnancy:

STAGE 1-Dose Identification: Phase 2a pharmacokinetic (PK) study. Using an intensive sampling approach, the following detailed PK information about three doses of daily oral PrEP in pregnancy will be collected: standard FTC/TDF dose (200mg/300mg, n=18), 150% standard dose (300mg/450mg, n=18), and 200% standard dose (400mg/600mg, n=18). Following a lead-in period-where participants receive PrEP for 14 days under direct observation to reach steady state concentrations-plasma, peripheral blood mononuclear cells (PBMC), and other specimens are collected over a 24-hour period to characterize key PK parameters. During pregnancy, two cycles will be performed (i.e., during the second and third trimester) at the assigned FTC/TDF dose. For all participants, this cycle will be repeated at 12 weeks postpartum using the standard FTC/TDF dose, providing a within-person non-pregnant comparator in the longitudinal assessment of bioequivalence. Standard dose FTC/TDF will be offered between periods of direct observation.

INTERMEDIARY STEP-Independent Review: Findings from the initial dose identification stage will be independently reviewed by the Study Monitoring Committee. Based on assessments of the PK, tolerability and preliminary safety data, the committee is expected to recommend an increased dosage of FTC/TDF (150% vs. 200% standard dose) for further investigation in Stage 2.

STAGE 2-Extended Safety Assessment: Phase 2b open-label randomized trial. In the second stage, the extended safety of increased dose PrEP that was identified via independent review will be assessed. Comparison of standard vs. increased FTC/TDF dosages via an open-label randomized trial of 112 pregnant women, allocated 1:1 will be done. Because safety is inextricably linked to adherence, direct observation will be used to confirm adherence, but extend the exposure period through the remainder of pregnancy. Maternal safety will be assessed using detailed medical histories, symptoms diaries, and routine laboratory screening. Information about fetal growth, birth outcomes, and infant growth will be collected; and assessment of maternal and infant bone mineral density will be done twice in the early postpartum period. Embedded in this second stage is population PK sampling (i.e., in plasma, PBMCs, dried blood spot (DBS), and cervicovaginal fluid) to inform models of FTC/TDF concentrations over the course of pregnancy, to be developed as part of this study (Aim 3). Again, following the period of directly observed PrEP at the assigned dose in pregnancy, standard dose FTC/TDF will be self-administered postpartum, in accordance with local HIV guidelines.

** In this record, only activities related to Stage 1 of the study are described. When this advances to Stage 2, a separate entry record in clinicaltrials.gov will be created. **

ELIGIBILITY:
Inclusion Criteria:

Maternal participants:

* Aged 16 years or older
* PrEP-eligible by local guidelines
* Pregnant with a viable singleton pregnancy of between 14 and 23 completed weeks of gestation (from 14 weeks + 0 days to 23 weeks + 6 days) by ultrasonography at study entry
* HIV-negative based on the study-specific screening algorithm
* Hepatitis B surface antigen (HBsAg)-negative
* Weight >35 kg
* Provided informed consent and expressed willingness to participate in study activities with their infants, including daily administration of oral PrEP under direct observation

Infant participants:

Infant participants enter the study with their mother as unborn infants. There are no specific eligibility criteria for infant participation otherwise. If an infant is deemed too ill to undergo study procedures, procedures necessary for clinical management may be prioritized.

Exclusion Criteria:

Maternal participants will not enter the study if any of the following conditions are identified during the screening process:

* Grade 2 or greater laboratory parameters for alanine transaminase (ALT) or aspartate aminotransferase (AST), hemoglobin (HB), and absolute neutrophil count (ANC).
* Estimated creatinine clearance (CrCl) 90 mL/min or below, using the Cockcroft-Gault formula.
* Known history or evidence of current significant disease process, including: hematological conditions, renal disease, unexplained bone fractures, environmental enteric dysfunction, or allergies/sensitivities to FTC/TDF.
* Other current significant or uncontrolled disease process (active or chronic), substance use, or social circumstances that, in the judgment of the site investigator, would make participation in the study inappropriate or unsafe.
* Fetuses with known or suspected major fetal anomaly, either from screening ultrasound or via medical record
* Intention to leave the study site's catchment area before scheduled study exit.
* Current use of prohibited medications
* Concurrent use of other biomedical HIV prevention interventions (vaginal ring, injectable PrEP, any investigational prevention product).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 54 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Tenofovir diphosphate (TFV-DP) in peripheral blood mononuclear cells (PBMCs) | Up to 20 weeks after delivery
  AUC of TFV-DP

SECONDARY OUTCOMES:
Maternal grade >/= 2 adverse events | Up to 20 weeks after delivery
  The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS Adverse Event Grading Table), will be used to measure safety.
  These include grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening) events. Relatedness of adverse events will be assessed by site teams as defined in the protocol.
Adverse pregnancy outcomes | At time of delivery
  This is a composite outcome that includes fetal death (spontaneous abortion or stillbirth), preterm birth (<37 weeks gestation), and small for gestational age (<10%tile birthweight for gestational age according to INTERGROWTH 21st standards)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chi, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill; Lynda Stranix-Chibanda, MBChB, MMed, Principal Investigator — University of Zimbabwe; Peter Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (2):
- Bwaila District Hospital, Lilongwe, Malawi
- Seke North CRS, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Supporting Information: ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT06435026/ICF_000.pdf